CLINICAL TRIAL: NCT04560608
Title: Elucidating the Symptomatic, Explanatory and Prognostic Characteristics of GERIAtric Patients Hospitalized for COVID-19
Acronym: GERIA-COVID
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2020/100; ar20-0087v0 (Other: CNIL)
Record Dates: First submitted 2020-09-08; First posted 2020-09-23 (Actual); Last update posted 2021-12-20 (Actual); Status verified 2021-12

CONDITIONS: Covid19
Keywords: elderly; coronavirus disease
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Statement :

* The emerging Coronavirus 2019 (COVID-19) disease, linked to the SARS-CoV-2 (severe acute respiratory syndrome coronavirus 2) pathogen, has been spreading worldwide since December 2019, affecting millions of people and causing hundreds of thousands of deaths, particularly among the elderly.
* The first epidemiological evidence available reveals a different expression of the disease in the elderly, associated with a high risk of delayed diagnosis and implementation of protective measures and a particularly high morbidity and mortality, especially among the frailest.
* To date, there is no effective model for predicting the severity of COVID-19 in an individual.

The investigators hypothesize that there are specificities of COVID-19 in the elderly, both etiological, diagnostic and prognostic, all of which are not yet known and understood.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalization in the Geriatric unit of the University Hospital (UH) of Angers from 15/03/2020 and until the closure of the COVID-19 geriatric sector

Exclusion Criteria:

* Opposition to the use of the information collected for research purposes.

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: All consecutive patients meeting the eligibility criteria over the study period.
Sampling Method: Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2020-03-15 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Medical history and co-morbidities | baseline
  listing of medical history and co-morbidities data provided by the physician and the family during hospitalization
The physical examination data, and reports of relevant investigations data provided by the physician and the family during hospitalization | baseline
  The demographic characteristics are age, sex, marital status, place of life, career, presence of un/formal assistance, …
Electrocardiography QT Interval | baseline
  all electrocardiograms performed during hospitalization
Number of different therapeutic classes | baseline
  Number of different therapeutic classes taken per day.
Comprehensive Geriatric Assessment (CGA) | baseline
  Comprehensive geriatric assessment (CGA) is defined as a multidisciplinary diagnostic and treatment process that identifies medical, psychosocial, and functional capabilities of an older adult in order to develop a coordinated plan to maximize overall health with aging. CGA is based on the premise that a systematic evaluation of frail older persons by a team of health professionals may identify a variety of treatable health problems and lead to better health outcomes.
Biological parameters | baseline
  Characterization of the COVID-19 impact on the biological parameters evaluated by blood test.
Medical imaging results | baseline
  Assessment of lesion extension (percent) with medical imaging results (thoracic scan)
Diagnosis of COVID-19 | baseline
  Recovery of the diagnosis method (PCR or thoracic scan)
Length of hospitalization | at the 3-month follow-up
Number of death from any cause | at the 3-month follow-up
Reports of relevant investigations data provided by the physician and the family during the two-month telephone follow-up | at the 3-month follow-up
  The demographic characteristics are age, sex, marital status, place of life, career, presence of un/formal assistance, …
Length of hospitalization | at the 12-month follow-up
Number of death from any cause | at the 12-month follow-up
Reports of relevant investigations data provided by the physician and the family during the two-month telephone follow-up | at the 12-month follow-up
  The demographic characteristics are age, sex, marital status, place of life, career, presence of un/formal assistance, …

CONTACTS AND LOCATIONS:
Overall Officials: Cédric ANNWEILER, MD, PhD, Principal Investigator — University Hospital, Angers
Locations (1):
- Angers University Hospital, Angers, France

REFERENCES:
- [Derived] Briere O, Otekpo M, Asfar M, Gautier J, Sacco G, Annweiler C; GERIA-COVID study group. Initial functional disability as a 1-year prognostic factor in geriatric patients hospitalized with SARS-CoV-2 infection. PLoS One. 2023 Jul 27;18(7):e0289297. doi: 10.1371/journal.pone.0289297. eCollection 2023. PMID 37498909